CLINICAL TRIAL: NCT06299280
Title: The Effect Of Dual-Task Training On Motor And Cognitive Performance In School-Age Children
Acronym: Dual-task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igdir University (Other)
Responsible Party: Principal Investigator, Sema Bugusan Oruc, Head of Physiotherapy and Rehabilitation Department, Igdir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Igdir180
Record Dates: First submitted 2024-02-27; First posted 2024-03-07 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Healthy; Child, Only
Keywords: Dual Task; School-age Children

STUDY DESIGN:
Intervention Model Description: randomised controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dual-task group (Experimental): Cognitive tasks will be given simultaneously while students exercise in physical education class.
  Interventions: Other: dual task training
- single-task group (Experimental): Students exercise in physical education class.
  Interventions: Other: single task training

INTERVENTIONS:
Other: dual task training — students will be given additional cognitive tasks while exercising in physical education class
  Arms: dual-task group
Other: single task training — students will exercise in physical education class, without additional cognitive tasks
  Arms: single-task group

SUMMARY:
The aim of the study is to investigate the effect of dual task training on performance in school-age children. Although studies on this subject in the world are limited, a comprehensive study on school-age children is needed.

MATERIAL AND METHOD:

* Evaluation will begin by applying demographic information and the Physical Activity Survey for Children.
* The evaluations to be made will primarily evaluate the child's performance on a single cognitive task in a supported sitting position on a chair, without a motor task.
* To evaluate single motor performance, a 2-minute walk test and a 30-second sit-stand test will be applied.
* Dual task evaluations will be carried out by adding a cognitive task while applying the 2-minute walk and 30-second sit-to-stand test.
* Walking speed will be evaluated with the 10m walk test.
* Balance parameter will be evaluated with functional reaching test.
* Using the Visual Analog Scale (VAS), participating children will be asked to score the difficulty of cognitive and motor performance as a number between 0 and 10.
* Walking speeds will be normalized by measuring lower extremity lengths.
* The children will be randomly divided into two groups and the study group will be given dual-task training by creating dual-task situations during the activities carried out in physical education classes.
* After 4 weeks, appropriate analyzes will be made with the data obtained as a result of the evaluations performed by the same evaluator.

As a result of this study, motor and cognitive performance in single-task conditions in typically developing children will be revealed. Additionally, changes in this performance will be detected in dual-task situations. The gains to be obtained as a result of the training will also reveal the importance of implementing dual task training in school-age children.

DETAILED DESCRIPTION:
Performing a cognitive task such as communicating while performing postural tasks such as walking is called dual task.

Attentional resources are divided into dual-task (DT) situations that are frequently experienced in daily life. Due to this division, the secondary task affects postural performance. DT states can be motor-motor, motor-cognitive, or cognitive-cognitive.

Humans, like other living creatures, are born, develop and learn in a multisensory field. Children encounter many dual-task (DT) situations in their daily, social and academic lives where they need to share limited attention resources. When attentional capacities are exceeded, performance of the postural task, cognitive task, or both may be impaired, causing DT confusion. DT confusion occurs more clearly in children, the elderly, and individuals with neurological involvement.The aim of the study is to investigate the effect of dual task training on performance in school-age children. Although studies on this subject in the world are limited, a comprehensive study on school-age children is needed.The physical activity level of the participants will be evaluated with the Physical Activity Questionnaire for Children (PAQ-C). There are two forms: PAQ-C, which evaluates the physical activity levels of primary school children between the ages of 8-12, and Physical Activity Questionnaire for Adolescents (PAQ-A), which evaluates the physical activity levels of students between the ages of 13-18. The answers to all questions except the last question in the survey are scored according to the frequency of the activity. Never gets 1 point, most often gets 5 points. In the last question, the answer does not have any points. The answer must be yes or no. A high result score indicates a high level of physical activity. A Turkish validity and reliability study was conducted.

MATERIAL AND METHOD:

* Evaluation will begin by applying demographic information and the Physical Activity Survey for Children.
* The evaluations to be made will primarily evaluate the child's performance on a single cognitive task in a supported sitting position on a chair, without a motor task.
* To evaluate single motor performance, a 2-minute walk test and a 30-second sit-stand test will be applied.
* Dual task evaluations will be carried out by adding a cognitive task while applying the 2-minute walk and 30-second sit-to-stand test.
* Walking speed will be evaluated with the 10m walk test.
* Balance parameter will be evaluated with functional reaching test.
* Using the Visual Analog Scale (VAS), participating children will be asked to score the difficulty of cognitive and motor performance as a number between 0 and 10.
* Walking speeds will be normalized by measuring lower extremity lengths.
* The children will be randomly divided into two groups and the study group will be given dual-task training by creating dual-task situations during the activities carried out in physical education classes.
* After 4 weeks, appropriate analyzes will be made with the data obtained as a result of the evaluations performed by the same evaluator.

As a result of this study, motor and cognitive performance in single-task conditions in typically developing children will be revealed. Additionally, changes in this performance will be detected in dual-task situations. The gains to be obtained as a result of the training will also reveal the importance of implementing dual task training in school-age children.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 7-15,
* Not having a chronic disease
* Volunteering to participate in the study and signing a consent form.

Exclusion Criteria

* Experiencing a health problem that will affect the musculoskeletal system in the last year,
* Having a condition that prevents participation in physical education class.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Physical Activity Questionnaire for Children (PAQ-C) | 5minutes
  There are two forms: PAQ-C, which evaluates the physical activity levels of primary school children between the ages of 8-12, and PAQ-A, which evaluates the physical activity levels of students between the ages of 13-18. The answers to all questions except the last question in the survey are scored according to the frequency of the activity. Never gets 1 point, most often gets 5 points. A high result score indicates a high level of physical activity. A Turkish validity and reliability study was conducted
Physical Activity Questionnaire for Adolescent (PAQ-A) | 5minutes
  There are two forms: PAQ-C, which evaluates the physical activity levels of primary school children between the ages of 8-12, and PAQ-A, which evaluates the physical activity levels of students between the ages of 13-18. The answers to all questions except the last question in the survey are scored according to the frequency of the activity. Never gets 1 point, most often gets 5 points. A high result score indicates a high level of physical activity. A Turkish validity and reliability study was conducted
Single cognitive task performance | 1minute
  Single cognitive task performance will measure with n-back in sitting
2-minute walk test | 4minutes
  2-minute walk test (single and dual-task conditions)
30-second sit-stand test | 2minutes
  30-second sit-stand test (single and dual-task conditions)
10m walk test. (single-task conditions) | 2minutes
  10m walk test will be aplied. 10-meter walking time will be recorded.
10m walk test. (dual-task conditions) | 2minutes
  10m walk test. 10-meter walking time with concurrent cognitive task will be recorded.
functional reaching test. | 1minute
  functional reaching test.(single and dual-task conditions)
Visual Analog Scale (VAS) | 1minute
  Visual Analog Scale (VAS) for motor and cognitive task. The higher the score indicates the difficulty of the task (0=simple task, 10: difficult almost cannot do)
lower extremity lengths assessment | 1minute
  lower extremity lengths assessment with tape measure

CONTACTS AND LOCATIONS:
Locations (1):
- Iğdır University, Iğdır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hagmann-von Arx P, Manicolo O, Lemola S, Grob A. Walking in School-Aged Children in a Dual-Task Paradigm Is Related to Age But Not to Cognition, Motor Behavior, Injuries, or Psychosocial Functioning. Front Psychol. 2016 Mar 10;7:352. doi: 10.3389/fpsyg.2016.00352. eCollection 2016. PMID 27014158
- [Background] Barutchu A, Toohey S, Shivdasani MN, Fifer JM, Crewther SG, Grayden DB, Paolini AG. Multisensory perception and attention in school-age children. J Exp Child Psychol. 2019 Apr;180:141-155. doi: 10.1016/j.jecp.2018.11.021. Epub 2019 Jan 14. PMID 30655099
- [Background] Anderson M, Bucks RS, Bayliss DM, Della Sala S. Effect of age on dual-task performance in children and adults. Mem Cognit. 2011 Oct;39(7):1241-52. doi: 10.3758/s13421-011-0099-7. PMID 21538179
- [Background] Saxena S, Cinar E, Majnemer A, Gagnon I. Does dual tasking ability change with age across childhood and adolescence? A systematic scoping review. Int J Dev Neurosci. 2017 May;58:35-49. doi: 10.1016/j.ijdevneu.2017.01.012. Epub 2017 Feb 3. PMID 28167051
- [Background] Rabaglietti E, De Lorenzo A, Brustio PR. The Role of Working Memory on Dual-Task Cost During Walking Performance in Childhood. Front Psychol. 2019 Jul 31;10:1754. doi: 10.3389/fpsyg.2019.01754. eCollection 2019. PMID 31417472